CLINICAL TRIAL: NCT03451227
Title: A Pilot Study to Investigate the Efficacy and Safety of Dexmedetomidine and Fentanyl Versus Midazolam and Remifentanil for Sedation in Patients Undergoing Ablation Procedures for Treatment of a Tachyarrhythmia
Brief Title: Dexmedetomidine and Fentanyl Versus Midazolam and Remifentanil for Sedation in Patients Undergoing Ablation Procedures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit eligible participants
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Manager Anesthesia Research, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 13-6972-B
Record Dates: First submitted 2017-11-30; First posted 2018-03-01 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Tachyarrhythmia
Keywords: Sedation, Analgesia
MeSH Terms: conditions — Tachycardia; Agnosia

STUDY DESIGN:
Intervention Model Description: This is a prospective, single blind, randomised controlled study looking at the feasibility of dexmedetomidine for sedation during ablation procedures at Toronto General Hospital.
Who Masked: Participant, Care Provider
Masking Description: Patients will be randomly allocated (computer generated) to receive either a dexmedetomidine infusion or a remifentanil infusion.
  The patient, interventional cardiologist and data analyser will be blinded to the drugs given. The anaesthesia care provider will not be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine Group (Experimental): The study drug dexmedetomidine (PrecedexTM) is supplied as dexmedetomidine HCL 200mcg/vial (100mcg/ml). This will be added to 98 ml 0.9% NaCl to achieve a concentration of 2mcg/ml and infused at 0.2-1mcg/kg/hour from the start of the case. The infusion rate will be commenced at 1mcg/kg/hour in those less than or equal to 65 years of age, and at 0.7mcg/kg/hr in those greater than 65 years of age, and then titrated based on the intraoperative sedation scores (to achieve a Sedation and Agitation scale (SAS) score of less than or equal to 4) and cardiovascular parameters (within 30% of baseline).
  Interventions: Drug: Dexmedetomidine group
- Remifentanil Group (Active Comparator): Remifentanil HCL will be infused at 0.01-0.2 mcg/kg/min titrated to sedation level (SAS less than or equal to 4) and cardiovascular parameters (within 30% of baseline)
  Interventions: Drug: Remifentanil Group

INTERVENTIONS:
Drug: Dexmedetomidine group — The study drug dexmedetomidine (PrecedexTM) will be infused at 0.2-1mcg/kg/hour from the start of the case. The dexmedetomidine infusion will stop at completion of the procedure.
  Arms: Dexmedetomidine Group
Drug: Remifentanil Group — Remifentanil HCL will be infused at 0.01-0.2 mcg/kg/min titrated to sedation level (SAS less than or equal to 4) and cardiovascular parameters (within 30% of baseline). The infusion will be stopped at the end of the procedure.
  Arms: Remifentanil Group

SUMMARY:
To evaluate the safety and efficacy of dexmedetomidine and compare this to a current technique commonly used at TGH for sedation in patients undergoing ablation procedures for atrial fibrillation (AF) and atrial flutter.

The investigators hypothesise that dexmedetomidine will be at least equivalent to, or more so, in terms of effectiveness and safety, when compared to midazolam and remifentanil for sedation during ablation procedures.

DETAILED DESCRIPTION:
The role of ablation for chronic persistent AF has been debated amongst cardiologists for some time, and there is increasing evidence that ablation may be superior to medical management. As populations age, the rate of AF is likely to increase and therefore the numbers of ablations performed for this arrhythmia will also be expected to increase.

Ablation procedures can vary in length from one to more than 6 hours in duration and require the patient to keep still so as not to influence the mapping procedure.

Options for anaesthesia care include a general anaesthetic or sedation. Several studies have evaluated the safety of sedation for ablation, using combinations of fentanyl, midazolam and propofol. These demonstrate that the ablation procedures are well tolerated under deep sedation.

Dexmedetomidine is an attractive potential agent for this role due to its favourable respiratory pharmacodynamics and good sedation profile. Dexmedetomidine is a short acting relatively specific alpha-2 receptor agonist (alpha 2: alpha 1 = 1300:1). It has been shown to have very little effect on respiratory parameters, even at high doses.In addition, it may offer some analgesic properties and therefore minimise the need for narcotic based agents. the investigators will compare dexmedetomidine infusion and fentanyl bolus with remifentanil infusion midazolam bolus.

ELIGIBILITY:
Inclusion Criteria:

* patients listed for an ablation procedure for treatment of atrial fibrillation or flutter at TGH requiring sedation provided by an anesthetist
* Valid consent

Exclusion Criteria:

* Baseline HR <40
* Baseline SBP < 80mmHg
* Baseline SBP > 180mmHg
* Second or third degree heart block unless pacemaker in situ
* Uncontrolled heart failure/severe LV dysfunction (Ejection fraction < 40%)
* Severe hepatic dysfunction (Transaminases greater than 2 times the upper limit of normal)
* Renal dysfunction: estimated GFR < 30ml/min, or requiring dialysis
* Allergy to any of the study drugs (dexmedetomidine, remifentanil, fentanyl, midazolam)
* Cognitive impairment precluding ability to tolerate sedation and comply with assessment methods
* Requirement for general anaesthetic for the procedure
* Pregnancy or breast feeding mothers
* Chronic use or addiction to opioids
* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Number of haemodynamic events requiring intervention | up to 24 hours
  a.Hypotension i. A decrease of 30% or more from baseline ii. Or absolute cut off values of
  1. SBP < 80mmHg
  2. DBP <40mmHg iii. Number of events and total dose of phenylephrine or ephedrine administered.
     b. Hypertension i. An increase in Systolic blood pressure 30% or more from baseline ii. Or an absolute cut off value of > 180mmHg iii. Total number of events c. Bradycardia i. A decrease of 30% or more from baseline ii. Or absolute cut off values of < 40bpm iii. Total number of events and total dose of glycopyrolate or atropine administered.
Number of respiratory events requiring intervention | up to 24 hours
  Respiratory events requiring intervention
  1. Respiratory rate < 6 breaths/min
  2. Airway obstruction requiring manual support
  3. Airway obstruction requiring guedel insertion
  4. Apnoea (cessation of respiration >10seconds)
  5. Hypoxia (saturations <90% for >20 seconds)

SECONDARY OUTCOMES:
Intraoperative pain scores | up to 24 hours
  1. VAS score (visual analog score). VAS is a simple assessment tool consisting of a 10 cm line with 0 on one end, representing no pain, and 10 on the other, representing the worst pain ever experienced, which a patient indicates so the clinician knows the severity of his or her pain. Pain scores using a VAS scale ranging from zero to ten will be recorded every 30 minutes
  2. Total amount of additional fentanyl used intraoperatively
Intraoperative sedation scores | up to 24 hours
  1. Sedation Agitation Scale (SAS) scale range from 1 to 7 will be recorded every 5 minutes. The SAS scale is outlined below with an optimal score of 4 for procedural sedation.
     Ref: Riker RR, Picard JT and Fraser GL. Prospective evaluation of the Sedation-Agitation Scale for adult critically ill patients. Critical Care Medicine 1999;27(7):1325-1329.
  2. Total amount of additional midazolam used intraoperatively
Patient satisfaction | up to 48 hours
  Assessed with the Iowa Satisfaction with Anaesthesia scale 24 hours post procedure b. Assessor blinded to technique c. To include direct questioning regarding the patients willingness to undergo the same procedure again using the same technique
  Iowa Satisfaction with Anaesthesia scale
  Ref: Dexter F, Aker J, Wright W. Development of a measure of patient satisfaction with monitored anaesthetic care: the Iowa Satisfaction with Anesthesia Scale. Anesthesiology 1997; 87: 865-73.
  Patient assessment
  1. I threw up or felt like throwing up
  2. I would have the same anaesthetic again
  3. I itched
  4. I felt relaxed
  5. I felt pain
  6. I felt safe
  7. I was too hot or cold
  8. I was satisfied with the anesthesia care
  9. I felt pain during the surgery
  10. I felt good
  11. I hurt
Recovery time | up to 24 hours
  Time from stopping infusion to a SAS score of ≥4
Length of stay in the recovery unit | up to 24 hours
  Total time spent in recovery until appropriate discharge criteria are met and patient is discharged to the ward
Analgesia requirements | up to 24 hours
  Quantity of opioids required i. Intraoperatively ii. In recovery iii. In the first 24 hours post op
Post operative nausea and vomiting (PONV) | up to 24 hours
  1. Subjective or objective evidence of PONV lasting > 30 mins
  2. Antiemetic therapy administered
Itch | up to 24 hours
  Any complaints of itch during the procedure and 24 hours post operatively

CONTACTS AND LOCATIONS:
Overall Officials: George Djaiani, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, Univerity health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verma A, Natale A. Should atrial fibrillation ablation be considered first-line therapy for some patients? Why atrial fibrillation ablation should be considered first-line therapy for some patients. Circulation. 2005 Aug 23;112(8):1214-22; discussion 1231. doi: 10.1161/CIRCULATIONAHA.104.478263. No abstract available. PMID 16116072
- [Background] Di Biase L, Santangeli P, Natale A. How to ablate long-standing persistent atrial fibrillation? Curr Opin Cardiol. 2013 Jan;28(1):26-35. doi: 10.1097/HCO.0b013e32835b59bb. PMID 23207492
- [Background] Cappato R, Calkins H, Chen SA, Davies W, Iesaka Y, Kalman J, Kim YH, Klein G, Natale A, Packer D, Skanes A, Ambrogi F, Biganzoli E. Updated worldwide survey on the methods, efficacy, and safety of catheter ablation for human atrial fibrillation. Circ Arrhythm Electrophysiol. 2010 Feb;3(1):32-8. doi: 10.1161/CIRCEP.109.859116. Epub 2009 Dec 7. PMID 19995881
- [Background] Drabek T, Nemec J. Anesthetic management of electrophysiological procedures for heart failure. Int Anesthesiol Clin. 2012 Summer;50(3):22-42. doi: 10.1097/AIA.0b013e3182603e95. PMID 22735718
- [Background] Di Biase L, Conti S, Mohanty P, Bai R, Sanchez J, Walton D, John A, Santangeli P, Elayi CS, Beheiry S, Gallinghouse GJ, Mohanty S, Horton R, Bailey S, Burkhardt JD, Natale A. General anesthesia reduces the prevalence of pulmonary vein reconnection during repeat ablation when compared with conscious sedation: results from a randomized study. Heart Rhythm. 2011 Mar;8(3):368-72. doi: 10.1016/j.hrthm.2010.10.043. Epub 2010 Nov 2. PMID 21055479
- [Background] Di Biase L, Saenz LC, Burkhardt DJ, Vacca M, Elayi CS, Barrett CD, Horton R, Bai R, Siu A, Fahmy TS, Patel D, Armaganijan L, Wu CT, Kai S, Ching CK, Phillips K, Schweikert RA, Cummings JE, Arruda M, Saliba WI, Dodig M, Natale A. Esophageal capsule endoscopy after radiofrequency catheter ablation for atrial fibrillation: documented higher risk of luminal esophageal damage with general anesthesia as compared with conscious sedation. Circ Arrhythm Electrophysiol. 2009 Apr;2(2):108-12. doi: 10.1161/CIRCEP.108.815266. Epub 2009 Feb 13. PMID 19808454
- [Background] Wutzler A, Rolf S, Huemer M, Parwani AS, Boldt LH, Herberger E, Hohenbichler K, Dietz R, Haverkamp W. Safety aspects of deep sedation during catheter ablation of atrial fibrillation. Pacing Clin Electrophysiol. 2012 Jan;35(1):38-43. doi: 10.1111/j.1540-8159.2011.03260.x. Epub 2011 Nov 6. PMID 22054234
- [Background] Kottkamp H, Hindricks G, Eitel C, Muller K, Siedziako A, Koch J, Anastasiou-Nana M, Varounis C, Arya A, Sommer P, Gaspar T, Piorkowski C, Dagres N. Deep sedation for catheter ablation of atrial fibrillation: a prospective study in 650 consecutive patients. J Cardiovasc Electrophysiol. 2011 Dec;22(12):1339-43. doi: 10.1111/j.1540-8167.2011.02120.x. Epub 2011 Jun 21. PMID 21692895
- [Background] Salukhe TV, Willems S, Drewitz I, Steven D, Hoffmann BA, Heitmann K, Rostock T. Propofol sedation administered by cardiologists without assisted ventilation for long cardiac interventions: an assessment of 1000 consecutive patients undergoing atrial fibrillation ablation. Europace. 2012 Mar;14(3):325-30. doi: 10.1093/europace/eur328. Epub 2011 Oct 23. PMID 22024600
- [Background] Bhananker SM, Posner KL, Cheney FW, Caplan RA, Lee LA, Domino KB. Injury and liability associated with monitored anesthesia care: a closed claims analysis. Anesthesiology. 2006 Feb;104(2):228-34. doi: 10.1097/00000542-200602000-00005. PMID 16436839
- [Background] Candiotti KA, Bergese SD, Bokesch PM, Feldman MA, Wisemandle W, Bekker AY; MAC Study Group. Monitored anesthesia care with dexmedetomidine: a prospective, randomized, double-blind, multicenter trial. Anesth Analg. 2010 Jan 1;110(1):47-56. doi: 10.1213/ane.0b013e3181ae0856. Epub 2009 Aug 27. PMID 19713256
- [Background] Khan ZP, Ferguson CN, Jones RM. alpha-2 and imidazoline receptor agonists. Their pharmacology and therapeutic role. Anaesthesia. 1999 Feb;54(2):146-65. doi: 10.1046/j.1365-2044.1999.00659.x. PMID 10215710
- [Background] Belleville JP, Ward DS, Bloor BC, Maze M. Effects of intravenous dexmedetomidine in humans. I. Sedation, ventilation, and metabolic rate. Anesthesiology. 1992 Dec;77(6):1125-33. doi: 10.1097/00000542-199212000-00013. PMID 1361310
- [Background] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460
- [Background] Ebert TJ, Hall JE, Barney JA, Uhrich TD, Colinco MD. The effects of increasing plasma concentrations of dexmedetomidine in humans. Anesthesiology. 2000 Aug;93(2):382-94. doi: 10.1097/00000542-200008000-00016. PMID 10910487
- [Background] Ryu JH, Lee SW, Lee JH, Lee EH, Do SH, Kim CS. Randomized double-blind study of remifentanil and dexmedetomidine for flexible bronchoscopy. Br J Anaesth. 2012 Mar;108(3):503-11. doi: 10.1093/bja/aer400. Epub 2011 Dec 15. PMID 22174346
- [Background] Arain SR, Ruehlow RM, Uhrich TD, Ebert TJ. The efficacy of dexmedetomidine versus morphine for postoperative analgesia after major inpatient surgery. Anesth Analg. 2004 Jan;98(1):153-158. doi: 10.1213/01.ANE.0000093225.39866.75. PMID 14693611
- [Background] Cortinez LI, Hsu YW, Sum-Ping ST, Young C, Keifer JC, Macleod D, Robertson KM, Wright DR, Moretti EW, Somma J. Dexmedetomidine pharmacodynamics: Part II: Crossover comparison of the analgesic effect of dexmedetomidine and remifentanil in healthy volunteers. Anesthesiology. 2004 Nov;101(5):1077-83. doi: 10.1097/00000542-200411000-00006. PMID 15505442
- [Background] Kaygusuz K, Gokce G, Gursoy S, Ayan S, Mimaroglu C, Gultekin Y. A comparison of sedation with dexmedetomidine or propofol during shockwave lithotripsy: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):114-9, table of contents. doi: 10.1213/01.ane.0000296453.75494.64. PMID 18165564
- [Background] Angst MS, Ramaswamy B, Davies MF, Maze M. Comparative analgesic and mental effects of increasing plasma concentrations of dexmedetomidine and alfentanil in humans. Anesthesiology. 2004 Sep;101(3):744-52. doi: 10.1097/00000542-200409000-00024. PMID 15329600
- [Background] Talke P, Li J, Jain U, Leung J, Drasner K, Hollenberg M, Mangano DT. Effects of perioperative dexmedetomidine infusion in patients undergoing vascular surgery. The Study of Perioperative Ischemia Research Group. Anesthesiology. 1995 Mar;82(3):620-33. doi: 10.1097/00000542-199503000-00003. PMID 7879930
- [Background] Arain SR, Ebert TJ. The efficacy, side effects, and recovery characteristics of dexmedetomidine versus propofol when used for intraoperative sedation. Anesth Analg. 2002 Aug;95(2):461-6, table of contents. doi: 10.1097/00000539-200208000-00042. PMID 12145072
- [Background] Hogue CW Jr, Talke P, Stein PK, Richardson C, Domitrovich PP, Sessler DI. Autonomic nervous system responses during sedative infusions of dexmedetomidine. Anesthesiology. 2002 Sep;97(3):592-8. doi: 10.1097/00000542-200209000-00012. PMID 12218525
- [Background] Venn M, Newman J, Grounds M. A phase II study to evaluate the efficacy of dexmedetomidine for sedation in the medical intensive care unit. Intensive Care Med. 2003 Feb;29(2):201-7. doi: 10.1007/s00134-002-1579-9. Epub 2002 Nov 22. PMID 12594584
- [Background] Jalowiecki P, Rudner R, Gonciarz M, Kawecki P, Petelenz M, Dziurdzik P. Sole use of dexmedetomidine has limited utility for conscious sedation during outpatient colonoscopy. Anesthesiology. 2005 Aug;103(2):269-73. doi: 10.1097/00000542-200508000-00009. PMID 16052108
- [Background] Hsu YW, Cortinez LI, Robertson KM, Keifer JC, Sum-Ping ST, Moretti EW, Young CC, Wright DR, Macleod DB, Somma J. Dexmedetomidine pharmacodynamics: part I: crossover comparison of the respiratory effects of dexmedetomidine and remifentanil in healthy volunteers. Anesthesiology. 2004 Nov;101(5):1066-76. doi: 10.1097/00000542-200411000-00005. PMID 15505441
- [Background] Alhashemi JA. Dexmedetomidine vs midazolam for monitored anaesthesia care during cataract surgery. Br J Anaesth. 2006 Jun;96(6):722-6. doi: 10.1093/bja/ael080. Epub 2006 Apr 4. PMID 16595611
- [Background] Vann MA, Ogunnaike BO, Joshi GP. Sedation and anesthesia care for ophthalmologic surgery during local/regional anesthesia. Anesthesiology. 2007 Sep;107(3):502-8. doi: 10.1097/01.anes.0000278996.01831.8d. PMID 17721254
- [Background] Cheung CW, Ying CL, Chiu WK, Wong GT, Ng KF, Irwin MG. A comparison of dexmedetomidine and midazolam for sedation in third molar surgery. Anaesthesia. 2007 Nov;62(11):1132-8. doi: 10.1111/j.1365-2044.2007.05230.x. PMID 17924894
- [Background] Sichrovsky TC, Mittal S, Steinberg JS. Dexmedetomidine sedation leading to refractory cardiogenic shock. Anesth Analg. 2008 Jun;106(6):1784-6. doi: 10.1213/ane.0b013e318172fafc. PMID 18499610
- [Background] McCutcheon CA, Orme RM, Scott DA, Davies MJ, McGlade DP. A comparison of dexmedetomidine versus conventional therapy for sedation and hemodynamic control during carotid endarterectomy performed under regional anesthesia. Anesth Analg. 2006 Mar;102(3):668-75. doi: 10.1213/01.ane.0000197777.62397.d5. PMID 16492813
- [Background] Rozet I, Muangman S, Vavilala MS, Lee LA, Souter MJ, Domino KJ, Slimp JC, Goodkin R, Lam AM. Clinical experience with dexmedetomidine for implantation of deep brain stimulators in Parkinson's disease. Anesth Analg. 2006 Nov;103(5):1224-8. doi: 10.1213/01.ane.0000239331.53085.94. PMID 17056959
- [Background] Okawa K, Ichinohe T, Kaneko Y. A comparison of propofol and dexmedetomidine for intravenous sedation: a randomized, crossover study of the effects on the central and autonomic nervous systems. Anesth Analg. 2010 Feb 1;110(2):415-8. doi: 10.1213/ANE.0b013e3181c88ba0. Epub 2009 Dec 10. PMID 20007736
- [Background] Tsai CJ, Chu KS, Chen TI, Lu DV, Wang HM, Lu IC. A comparison of the effectiveness of dexmedetomidine versus propofol target-controlled infusion for sedation during fibreoptic nasotracheal intubation. Anaesthesia. 2010 Mar;65(3):254-9. doi: 10.1111/j.1365-2044.2009.06226.x. Epub 2010 Jan 22. PMID 20105150
- [Background] Dupanovic M, Lakkireddy D, Emert MP, Krebill R. Utility of dexmedetomidine in sedation for radiofrequency ablation of atrial fibrillation. J Perianesth Nurs. 2013 Jun;28(3):144-50. doi: 10.1016/j.jopan.2012.10.005. PMID 23711310
- [Background] Prachanpanich N, Apinyachon W, Ittichaikulthol W, Moontripakdi O, Jitaree A. A comparison of dexmedetomidine and propofol in Patients undergoing electrophysiology study. J Med Assoc Thai. 2013 Mar;96(3):307-11. PMID 23539933
- [Background] Riker RR, Picard JT, Fraser GL. Prospective evaluation of the Sedation-Agitation Scale for adult critically ill patients. Crit Care Med. 1999 Jul;27(7):1325-9. doi: 10.1097/00003246-199907000-00022. PMID 10446827
- [Background] Dexter F, Aker J, Wright WA. Development of a measure of patient satisfaction with monitored anesthesia care: the Iowa Satisfaction with Anesthesia Scale. Anesthesiology. 1997 Oct;87(4):865-73. doi: 10.1097/00000542-199710000-00021. PMID 9357889